CLINICAL TRIAL: NCT03516695
Title: RadioEmbolization for the ADvancement of Y90 Glass Microspheres Registry
Acronym: READ90Y
Status: Terminated | Type: Observational
Why Stopped: due to Sponsor's ongoing and upcoming projects and overall research priorities
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BTG-007509-01
Record Dates: First submitted 2018-03-22; First posted 2018-05-04 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Liver Cancer
Keywords: Registry; Liver Cancers; HCC; Dosimetry; Simplicit90Y™; TheraSphere®
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TheraSphere® — Intra-arterial Yttrium-90 glass microspheres

SUMMARY:
This study is a non-interventional, observational, prospective, and global participant data registry. The study will collect effectiveness and safety data from approximately 1000 participants with liver cancers treated with TheraSphere® in a real-life setting from multiple centers globally. The absorbed dose to tumor and normal tissue will be calculated using the Simplicit90Y™ software in the subgroup of hepatocellular carcinoma (HCC) participants.

DETAILED DESCRIPTION:
This study is a non-interventional, observational, prospective and global participant data registry.

Approximately 1000 participants with liver cancers who are treated with TheraSphere® will be enrolled.

Data regarding participant and treatment characteristics (TheraSphere® and other anti-cancer treatments) will be collected within a 12-month period post TheraSphere® administration to:

* Assess treatment effectiveness and safety in a real-life administration setting
* Identify prognostic and predictive factors for liver cancer participants receiving TheraSphere® treatment

Data for dosimetry determination will be collected on approximately 300 HCC participants to assess:

* Technetium-99m Macroaggregated albumin (99mTc-MAA) normal tissue and tumor Absorbed Dose using pre-procedural Single Proton Emission Computed Tomography/ Computed Tomography (SPECT/CT)
* Yttrium-90 and isotopes (Y90) normal tissue and tumor Absorbed Dose using post-procedural PET/CT (or equivalent for Asia) scans

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥ 18 years of age
2. Participant has confirmed liver cancer
3. Participant is able to provide informed consent according to local requirements/law
4. Participant has a life expectancy of ≥ 3 months
5. Participant is scheduled to receive TheraSphere® treatment

Exclusion Criteria:

1. Participant who has previously received Y90 microspheres
2. Participant who has consented to participate in a BTG-sponsored clinical study that includes TheraSphere® treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with liver cancer for whom treatment with TheraSphere® has been prescribed and who meet all study eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of TheraSphere® treatment in participants with liver cancers in a real-life setting | 12 months follow up post last TheraSphere® treatment
  Tumor response to TheraSphere® treatment will be assessed using Modified Response Evaluation Criteria in Solid Tumors (mRECIST) or Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 depending on tumor type.

SECONDARY OUTCOMES:
Serious adverse events | 6 months follow up post last TheraSphere® treatment
  Serious adverse events assessed as related or possibly related to TheraSphere®.
Adverse events of interest | 6 months follow up post last TheraSphere® treatment
  Specific adverse events assessed as related or possibly related to TheraSphere®, comprising of any of the following events: fatigue, pain, nausea, ascites, lymphopenia, hyperbilirubinemia, hypoalbuminemia.
TheraSphere® Dosimetry in the subgroup of HCC participants | From up to 30 days until the date of TheraSphere® Treatment and Baseline
  Dose absorbed to normal tissue and tumor, using the pre TheraSphere® 99mTc-MAA SPECT/CT, will be examined and compared to post TheraSphere® Y90 PET/CT (or equivalent in Asia) using the Simplicit90Y™ software.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Lencioni, MD, Principal Investigator — University of Miami (previously known affiliation)
Locations (8):
- United States (7):
  - UCLA, Los Angeles, California
  - University of Miami, Coral Gables, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Allina Health System Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - New York University School of Medicine, New York, New York
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- See also: Sponsor Website — http://www.btgplc.com